CLINICAL TRIAL: NCT07276516
Title: The Investigation of the Effects of Academic Stress and Burnout on Musculoskeletal Disorders in Academicians
Brief Title: Psychosocial Factors Related to Musculoskeletal Disorders in Academicians
Acronym: MSDs
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, ERDİ KAYABINAR, Assistant Professor, University of Yalova
Other Study IDs: 2024/292
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Musculoskeletal Disorders
Keywords: musculoskeletal disorders; academic stress; burnout; work-life balance
MeSH Terms: conditions — Musculoskeletal Diseases; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Academicians: Academicans with muscoloskeletal disorders

SUMMARY:
the prevalence of occupational stress and burnout is very high among academicians. Previous studies examining MSDs in academicians have focused more on physical factors such as physical activity levels and ergonomics, while interest in psychosocial factors has been limited. To our knowledge, there is no study in the literature that evaluates both MSDs, work stress, and burnout in academicians. Therefore, our study aims to investigate the relationship between MSDs and academic stress, burnout, and work-life balance among academicians.

DETAILED DESCRIPTION:
The study aims to investigate psychosocial factors such as academic stress and burnout, which are thought to influence musculoskeletal disorders among academics. As part of the research, data will be collected through questionnaires from volunteer academics at a selected university who have at least six months of teaching experience at the institution. The questionnaire will gather information on musculoskeletal pain, demographic characteristics, stress levels, burnout levels, and work-life balance. After entering the data into the SPSS software, statistical analysis will be conducted. Categorical variables will be presented as numbers (percentages), and numerical variables will be reported as means and standard deviations. To assess correlations, Spearman or Pearson correlation tests and regression analyses will be used. The Chi-square test will be used to compare categorical variables between male and female academics, while the independent samples t-test will be applied for numerical variables if normality is assumed; otherwise, the Mann-Whitney U test will be used. The Shapiro-Wilk test will be conducted to assess the normality of the data. A significance level of p<0.005 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate,
* having worked as academic staff at Yalova University for the past six months,
* being able to understand and speak Turkish

Exclusion Criteria:

* who wished to withdraw from the study,
* those with a history of fracture or soft tissue injury in any body region within the past 12 months,
* congenital spinal disorders, scoliosis, rheumatoid diseases, cancer, surgery, chronic internal organ pain, long-term use of analgesic or psychiatric medications, - those working in departments without students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Academicians who worked as academic staff at Yalova University for the past six months
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
The Extended Nordic Musculoskeletal Questionnaire | All participants will be assessed only once.
  Dawson and colleagues developed an extended version of the Nordic Musculoskeletal Questionnaire to obtain more detailed data on the prevalence and impact of musculoskeletal disorders. It includes general questions about the history of problems in nine body regions, such as the neck, upper back, shoulders, elbows, hands/arms, lower back, hips, knees, and feet/ankles. The questionnaire was provided along with a body diagram to help participants indicate areas of pain or discomfort. The response options are limited to "yes" and "no." A Turkish cultural adaptation and validity study of the questionnaire has been conducted.
University Academic Staff Work Stress Scale | All participants will be assessed only once.
  University Academic Staff Work Stress Scale, developed by Balcı in 1992 and validated for reliability and validity, was used. The scale contains 24 items. The total scale score ranges from 0 to 120, with higher scores indicating lower job satisfaction. The questionnaire has high validity and reliability.
The Maslach Burnout Inventory | All participants will be assessed only once.
  The Maslach Burnout Inventory was developed by Maslach and Jackson in 1981. The inventory has also been validated and tested for reliability for use in Turkish among academicians. The inventory consists of 22 items and assesses burnout across three subscales: emotional exhaustion, depersonalization, and personal accomplishment. The emotional exhaustion subscale includes nine items related to fatigue, boredom, and reduced emotional energy. The depersonalization subscale consists of five items concerning detached or impersonal behavior toward care and service recipients. The personal accomplishment subscale comprises eight items and reflects an individual's sense of competence and achievement. Items on the scale are rated on a Likert scale from 0 to 6. Separate scores were obtained for each of the three subscales. High scores on the emotional exhaustion or depersonalization subscales, or low scores on the personal accomplishment subscale, indicate a high level of burnout.

SECONDARY OUTCOMES:
Work-Life Balance Scale | All participants will be assessed only once.
  The scale, developed and tested for reliability by Taşdelen-Karçkay and Bakalım, evaluates the balance between work and life. It consists of 8 items rated on a 7-point Likert scale, with each item scored from "Strongly Disagree -1-" to "Strongly Agree -7-." Low scores indicate a disruption in work-life balance.

CONTACTS AND LOCATIONS:
Overall Officials: Erdi KAYABINAR, PhD, Principal Investigator — University of Yalova
Locations (1):
- University of Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researchers do not plan to share the data due to concerns about data confidentiality.

REFERENCES:
- [Background] Taşdelen-Karçkay A, Bakalım OJAJoCD. The mediating effect of work-life balance on the relationship between work-family conflict and life satisfaction. 2017;26(1):3-13.
- [Background] Balcı A. ÜNİVERSİTE ÖĞRETİM ELEMANININ İŞ STRESİ ÖLÇEĞİ. Ankara University Journal of Faculty of Educational Sciences (JFES). 1992;26(1):315-34.
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Abbak Y, Toprak E, Çelebi MJUTEKED. A STUDY OF CAREER BARRIERS AND OCCUPATIONAL BURNOUT LEVELS OF ACADEMICIANS IN EDUCATION FACULTY ACCORDING TO VARIOUS DEMOGRAPHIC VARIABLES. 2024;13(2):735-59.
- [Background] Maslach C, Jackson SEJJoob. The measurement of experienced burnout. 1981;2(2):99-113.
- [Background] Bongers PM, de Winter CR, Kompier MA, Hildebrandt VH. Psychosocial factors at work and musculoskeletal disease. Scand J Work Environ Health. 1993 Oct;19(5):297-312. doi: 10.5271/sjweh.1470. PMID 8296178
- [Background] Ozdinc S, Kayabinar E, Ozen T, Turan FN, Yilmaz S. Musculoskeletal problems in academicians and related factors in Turkey. J Back Musculoskelet Rehabil. 2019;32(6):833-839. doi: 10.3233/BMR-181171. PMID 31403936
- [Background] Ayaz J, Ghaffar T, Iqbal A, Arshad S, Aroofa H, Nasir M, et al. Musculoskeletal Disorders Risk Factors among Faculty Members of Academic Institute: Musculoskeletal Disorders Risk Factors. Pakistan Journal of Health Sciences. 2023.